CLINICAL TRIAL: NCT01814631
Title: Prospective Comparison of Two EUS Processors for Imaging of the Pancreas
Brief Title: Endoscopic Ultrasound (EUS) Processor Comparison
Status: Withdrawn | Type: Observational
Why Stopped: Closed at PI discretion
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 409829
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Pancreatitis; Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatitis; Pancreatic Neoplasms | interventions — Pharmaceutical Solutions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aloka: image quality and resolution
  Interventions: Other: image quality and resolution

INTERVENTIONS:
Other: image quality and resolution — Image quality and resolution will be viewed using Aloka processor
  Other Names: Aloka
Other: image quality and resolution — image quality and resolution will be viewed on the EU-me2
  Other Names: EU-me2

SUMMARY:
The primary objective for this study is to compare the image quality of two endoscopic ultrasound (EUS) processors used for imaging of the pancreas. Processor images are used to make a correct clinical diagnosis and higher quality imaging is related to more accurate results. Patient care may be improved due to the information collected as part of this study.

The quality of imaging is of utmost importance for diagnosing early neoplasms in the pancreas and diseases such as chronic pancreatitis. Image quality is dictated by two factors: image resolution and depth of penetration. Good imaging enables diagnosis of early stage disease and thereby facilitates early treatment.

DETAILED DESCRIPTION:
The endoscope is usually connected to a processor that generates an image which is viewed on a monitor. At FH, we use a processor called Aloka 10. A new processor is being developed by Olympus Corporation called EU-ME 2. This new processor is FDA approved, but has not been launched commercially yet. It has been loaned to FH for evaluation. We would like to evaluate this processor in an objective manner and hence the request for study approval.

In this study, the endoscopy during the procedure will be attached to two different processors and images will be generated. The choice of which processor will be used first will be at the discretion of the Endoscopist. This does not require removal and reintroduction of the endoscope into the patient at two occasions. Only the connector will be switched to a different processor. So there is negligible risk to the patient.

The time required for research activities will be between 5-10 minutes. Both processors will be set up in the procedure room for the duration of this study.

The physician will then document the depth of penetration of the image (the farthest structure seen) and image resolution (evaluating the pancreas for subtle abnormalities). Both processors will be used for each patient. The scores for each processor will be documented to a procedure log, using the primary endpoint described above. The CRF will not have any patient information. Images viewed by the physician at the time of procedure will not be saved or recorded as part of this study..

EUS will be performed in the standard fashion by one of the experienced endosonographers in the unit. Once the EUS is complete, the procedure will be stopped and the echoendoscope withdrawn from the patient.

Patients will then be transported to the recovery area for observation as per standard policy. After appropriate observations are deemed satisfactory, patients will be discharged as per unit policy.

ELIGIBILITY:
Inclusion Criteria:

All patients referred to Florida Hospital Endoscopy Unit for assessment of pancreas will be included.

Exclusion Criteria:

Age <19 years Unable to safely undergo EUS for any reason

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients referred to Florida Hospital Endoscopy Unit for assessment of pancreas will be included.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
image quality | up to 2 months
  The primary endpoint of the study is to compare processors by assessing image resolution and depth of penetration. This will be accomplished using a objective scoring system assigning one point for each structure visualized. This score will range from 0 to a maximum of 9.

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No